CLINICAL TRIAL: NCT03477838
Title: A Pharmacist-driven Continuous Glucose Monitoring Program for Advanced Diabetes Management in an Uninsured Population
Brief Title: Pharmacist-driven CGM Use in the Uninsured Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM20012049
Record Dates: First submitted 2018-03-19; First posted 2018-03-26 (Actual); Results first posted 2021-02-05 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-01

CONDITIONS: Diabetes Mellitus
Keywords: continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- CGM Intervention arm (Experimental): Patients eligible for care at the free clinic with diabetes and A1c greater than 8% on insulin therapy will be identified for CGM use.
  Interventions: Device: FreeStyle LibrePro CGM

INTERVENTIONS:
Device: FreeStyle LibrePro CGM — a professional CGM device will be worn by the participant for up to 14 days

SUMMARY:
This is a pilot study. The purpose is to (1) provide access to continuous glucose monitoring (CGM) to patients (purchased through a grant) and (2) systematically record and analyze the results of the glucose monitoring by the clinical pharmacists at the clinic.

ELIGIBILITY:
Inclusion Criteria:

1. adult 18 years of age or older
2. diagnosis of Type 1 or Type 2 diabetes
3. A1c greater than 8%
4. prescribed basal insulin plus either prandial insulin or a glucagon-like peptide-1 (GLP-1) receptor agonist

Exclusion Criteria:

1. pregnant or breast-feeding
2. on dialysis
3. not appropriate for CGM use based on clinical judgment by the investigators
4. patients with limited English proficiency

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evan Sisson, PharmD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CGM Intervention Arm
Started | 28
Completed | 14
Not Completed | 14
Not completed — Lost to Follow-up | 14

BASELINE CHARACTERISTICS:
Arm/Group | CGM Intervention Arm
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] — Age was only collected on part of the study population. Population: Age data was not collected from all participants.
  years
    number analyzed (Participants) | 13
    (all) | 68 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Change in A1c
Description: Change in A1c will be used to assess glycemic control
Time Frame: Baseline to week 12
Measure: Mean (Standard Deviation); unit: percent of hemoglobin
Arm/Group | CGM Intervention Arm
Number analyzed (Participants) | 14
percent of hemoglobin | -0.74 (1.6)

2. Secondary Outcome: Medication Changes
Description: Data will be collected on what medication changes are made (changes in types of medications and doses)
Time Frame: Baseline to week 12
Measure: Mean (Standard Deviation); unit: number of medication changes
Arm/Group | CGM Intervention Arm
Number analyzed (Participants) | 14
number of medication changes | 1.83 (0.5)

3. Secondary Outcome: Glycemic Variability
Description: Data collected by the CGM, such as time-in-therapeutic range, will be evaluated to assess glycemic variability during the 14 day period of wearing the CGM
Time Frame: Baseline to week 12
Measure: Mean (Standard Deviation); unit: percent time in range
Arm/Group | CGM Intervention Arm
Number analyzed (Participants) | 14
percent time in range
  Time in Therapeutic goal | -3.17 (23.5)
  Time in Hypoglycemia | 2.58 (13.7)
  Time in Hyperglycemia | 1.5 (30.4)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | CGM Intervention Arm
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2018-03-11): https://cdn.clinicaltrials.gov/large-docs/38/NCT03477838/Prot_000.pdf